CLINICAL TRIAL: NCT01623180
Title: A Prospective Randomized Comparison of the BioFreedom Biolimus A9 Drug Coated Stent Versus the Gazelle Bare Metal Stent in Patients With High Risk of Bleeding.
Brief Title: A Randomized Clinical Evaluation of the BioFreedom™ Stent
Acronym: Leaders Free
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biosensors Europe SA (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12EU01
Record Dates: First submitted 2012-06-05; First posted 2012-06-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Stable Angina; Ischemic Heart Disease Silent; ST Elevation (STEMI) and Non-ST Elevation (NSTEMI) Myocardial Infarction; In-stent Coronary Artery Restenosis; Bleeding
Keywords: DES; coronary stent; bare metal stent; high bleeding; MI; angina
MeSH Terms: conditions — Angina, Stable; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Myocardial Infarction; Hemorrhage; Angina Pectoris | interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BioFreedom™ Drug Coated Stent (DCS) (Experimental): BA9 drug coated stent implantation for improving coronary luminal diameter in patients with de novo lesions in native coronary arteries with a reference vessel diameter between 2.25 mm and 4.0 mm.
  Interventions: Device: Biofreedom™ Drug Coated Stent (DCS)
- Gazelle™ Bare Metal Coronary Stent (BMS) (Active Comparator): GAZELLE™ bare metal stent implantation for improving coronary luminal diameter in patients with de novo lesions in native coronary arteries with a reference vessel diameter between 2.25 and 4.0 mm.
  Interventions: Device: Gazelle™ Bare Metal Coronary Stent (BMS)

INTERVENTIONS:
Device: Biofreedom™ Drug Coated Stent (DCS) — Biofreedom DCS implantation in high risk bleeding patients followed by 1 month DAPT
  Other Names: Drug coated stent
  Arms: BioFreedom™ Drug Coated Stent (DCS)
Device: Gazelle™ Bare Metal Coronary Stent (BMS) — Gazelle BMS implantation in high risk bleeding patients followed by 1 month DAPT
  Arms: Gazelle™ Bare Metal Coronary Stent (BMS)

SUMMARY:
The purpose of this study is to demonstrate that a BioFreedom™ Drug Coated Stent is non-inferior to a bare metal stent at one year as measured by the composite safety endpoint of cardiovascular death, myocardial infarction and definite/probable stent thrombosis, and that its efficacy is superior to a bare metal stent as measured by clinically driven TLR at one year.

ELIGIBILITY:
Inclusion Criteria:

* Any indication for PCI-S in patients deemed at high risk for bleeding and candidates for 1 month DAPT. This includes candidates with stable angina, silent ischemia, ACS (STEMI and non-STEMI), non-native lesions and in-stent restenosis. Patients must provide written informed consent.

Exclusion Criteria:

1. Pregnancy
2. Patients expected not to comply with 1 month DAPT
3. Patients requiring a planned staged PCI procedure more than one week after the index procedure
4. Procedure planned to require non-study stents, or stand alone POBA or stand-alone atherectomy
5. Active bleeding at the time of inclusion
6. Reference vessel diameter <2.25 - >4.0mm
7. Cardiogenic shock
8. Compliance with long-term single anti-platelet therapy unlikely
9. A known hypersensitivity or contraindication to aspirin, clopidogrel (or prasugrel, or ticagrelor if applicable), stainless steel, Biolimus A9 or a sensitivity to contrast media, which cannot be adequately pre-medicated.
10. Participation in another clinical trial (12 months after index procedure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2456 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-05 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Composite Safety Endpoint | one year
  Composite of cardiac death, myocardial infarction and definite/probable stent thrombosis at one year
Primary Efficacy Endpoint | one year
  The incidence of clinically driven target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Philip Urban, MD, Principal Investigator — Hôpital de la Tour
Locations (1):
- Hôpital de la Tour, Meyrin, Switzerland

REFERENCES:
- [Derived] Campos CM, Mehran R, Capodanno D, Owen R, Windecker S, Varenne O, Stone GW, Valgimigli M, Hajjar LA, Kalil Filho R, Oldroyd K, Morice MC, Urban P, Abizaid A. Risk Burden of Cancer in Patients Treated With Abbreviated Dual Antiplatelet Therapy After PCI: Analysis of Multicenter Controlled High-Bleeding Risk Trials. Circ Cardiovasc Interv. 2024 Apr;17(4):e013000. doi: 10.1161/CIRCINTERVENTIONS.122.013000. Epub 2024 Apr 16. PMID 38626080
- [Derived] Richardt G, Maillard L, Nazzaro MS, Abdel-Wahab M, Carrie D, Iniguez A, Garot P, Abdellaoui M, Morice MC, Foley D, Copt S, Stoll HP, Urban P. Polymer-free drug-coated coronary stents in diabetic patients at high bleeding risk: a pre-specified sub-study of the LEADERS FREE trial. Clin Res Cardiol. 2019 Jan;108(1):31-38. doi: 10.1007/s00392-018-1308-1. Epub 2018 Jun 27. PMID 29951803
- [Derived] Carrie D, Menown I, Oldroyd K, Copt S, Talwar S, Maillard L, Morice MC, Teik LS, Lang I, Urban P. Safety and Efficacy of Polymer-Free Biolimus A9-Coated Versus Bare-Metal Stents in Orally Anticoagulated Patients: 2-Year Results of the LEADERS FREE Oral Anticoagulation Substudy. JACC Cardiovasc Interv. 2017 Aug 28;10(16):1633-1642. doi: 10.1016/j.jcin.2017.05.033. PMID 28838473
- [Derived] Garot P, Morice MC, Tresukosol D, Pocock SJ, Meredith IT, Abizaid A, Carrie D, Naber C, Iniguez A, Talwar S, Menown IBA, Christiansen EH, Gregson J, Copt S, Hovasse T, Lurz P, Maillard L, Krackhardt F, Ong P, Byrne J, Redwood S, Windhovel U, Greene S, Stoll HP, Urban P; LEADERS FREE Investigators. 2-Year Outcomes of High Bleeding Risk Patients After Polymer-Free Drug-Coated Stents. J Am Coll Cardiol. 2017 Jan 17;69(2):162-171. doi: 10.1016/j.jacc.2016.10.009. Epub 2016 Oct 30. PMID 27806919
- [Derived] Urban P, Meredith IT, Abizaid A, Pocock SJ, Carrie D, Naber C, Lipiecki J, Richardt G, Iniguez A, Brunel P, Valdes-Chavarri M, Garot P, Talwar S, Berland J, Abdellaoui M, Eberli F, Oldroyd K, Zambahari R, Gregson J, Greene S, Stoll HP, Morice MC; LEADERS FREE Investigators. Polymer-free Drug-Coated Coronary Stents in Patients at High Bleeding Risk. N Engl J Med. 2015 Nov 19;373(21):2038-47. doi: 10.1056/NEJMoa1503943. Epub 2015 Oct 14. PMID 26466021
- [Derived] Urban P, Abizaid A, Chevalier B, Greene S, Meredith I, Morice MC, Pocock S. Rationale and design of the LEADERS FREE trial: A randomized double-blind comparison of the BioFreedom drug-coated stent vs the Gazelle bare metal stent in patients at high bleeding risk using a short (1 month) course of dual antiplatelet therapy. Am Heart J. 2013 May;165(5):704-9. doi: 10.1016/j.ahj.2013.01.008. Epub 2013 Feb 19. PMID 23622906